CLINICAL TRIAL: NCT03461861
Title: Network-Level Mechanisms for Preclinical Alzheimer's Disease Development
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Yang Wang, Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRO00031146; R21AG056882-01 (NIH)
Record Dates: First submitted 2018-02-26; First posted 2018-03-12 (Actual); Results first posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: APOE 4
Keywords: Healthy; Adult; Normal Memory; APOE 4; Brain; Magnetic Resonance Imaging; MRI; Alzheimer's disease; Hippocampus; Genetic testing; Dementia; AGB101
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled crossover study in which a low dose of AGB101 (220mg QD) or placebo will be administered to 50 healthy 55-75-year-old subjects, with the order of treatments counterbalanced in a within-subject crossover design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- AGB101 220 mg, then Placebo (Experimental): AGB101 220 mg/day capsule, once daily dosing for 2 weeks. After a 4 week washout, to be followed by Placebo, given as a capsule, once daily dosing for 2 weeks.
  Interventions: Drug: AGB101 220 mg; Other: Placebo
- Placebo, then AGB101 220 mg (Experimental): Placebo, given as a capsule, once daily for 2 weeks. After a 4 week washout, to be followed by AGB101 220 mg/day capsule, once daily dosing for 2 weeks.
  Interventions: Drug: AGB101 220 mg; Other: Placebo

INTERVENTIONS:
Drug: AGB101 220 mg — AGB101 oral dose of 220 mg/day capsule, given as once-daily dosing.
Other: Placebo — Placebo, oral capsule given once-daily.

SUMMARY:
The purpose of this project is to test the hypothesis that AGB101 low dose levetiracetam extended release formulation can reduce abnormal hyperfunctional activity in the hippocampus in normal, healthy adults. The investigators will compare the functional connectivity results after taking AGB101 or placebo.

DETAILED DESCRIPTION:
In this study the investigators want to find out whether the use of a perturbation, such as AGB101 low dose of levetiracetam extended release formulation, in healthy adults can reduce abnormal hippocampal network activity. The investigators also want to study whether this low dose of LEV can improve memory function.

Generic levetiracetam is a type of drug called an anti-epileptic or anti-seizure medication. It is FDA approved worldwide for adults and children as young as one month with seizures. It is a generic drug used in long-term epilepsy treatment. It is relatively safe and has an acceptable side-effect profile.

AGB101 has been developed as a novel extended release formulation of low dose levetiracetam (below clinically marketed doses for epilepsy) for slowing the progression of amnestic mild cognitive impairment.

It is known that age and the APOE 4 gene are important risk factors for late-onset Alzheimer's disease. Further studies have shown that cognitively normal, older adults have more hyperfunctional brain network activity, increased alpha beta accumulation, decreased memory function, and decreased brain volume, which is consistent with Alzheimer's disease patterns.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English
* At least eight (8) years of education
* Geriatric Depression Scale (GDS) (62) score < 6
* Hachinski Ischemic Score ≤ 4
* Normal general cognitive function as well as 1) normal memory function, documented by MOCA score of 23 or greater, and a RBANS Delayed Memory Index score of 85 or greater.

Exclusion Criteria:

* Neurological disease, such as Parkinson's disease, multi-infarct dementia, Huntington's disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, or a history of significant head trauma or known structural brain abnormalities
* Major psychiatric disease or chronic unstable medical conditions
* History of drug abuse
* History of alcohol abuse (4 or greater drinks per day on average)
* Unable to complete MRI scans (no Pacemaker/Defibrillator)
* Known clinically significant abnormalities in B12 or thyroid function tests
* End Stage Renal Disease (ESRD)
* Hemodialysis (HD)

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yang Wang, PhD, Principal Investigator — The Medical College of Wisconsin
Locations (1):
- Froedtert & The Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reiman EM, Chen K, Alexander GE, Caselli RJ, Bandy D, Osborne D, Saunders AM, Hardy J. Functional brain abnormalities in young adults at genetic risk for late-onset Alzheimer's dementia. Proc Natl Acad Sci U S A. 2004 Jan 6;101(1):284-9. doi: 10.1073/pnas.2635903100. Epub 2003 Dec 19. PMID 14688411
- [Background] Filippini N, MacIntosh BJ, Hough MG, Goodwin GM, Frisoni GB, Smith SM, Matthews PM, Beckmann CF, Mackay CE. Distinct patterns of brain activity in young carriers of the APOE-epsilon4 allele. Proc Natl Acad Sci U S A. 2009 Apr 28;106(17):7209-14. doi: 10.1073/pnas.0811879106. Epub 2009 Apr 8. PMID 19357304
- [Background] Sheline YI, Raichle ME, Snyder AZ, Morris JC, Head D, Wang S, Mintun MA. Amyloid plaques disrupt resting state default mode network connectivity in cognitively normal elderly. Biol Psychiatry. 2010 Mar 15;67(6):584-7. doi: 10.1016/j.biopsych.2009.08.024. Epub 2009 Oct 14. PMID 19833321
- [Background] Li W, Antuono PG, Xie C, Chen G, Jones JL, Ward BD, Singh SP, Franczak MB, Goveas JS, Li SJ. Aberrant functional connectivity in Papez circuit correlates with memory performance in cognitively intact middle-aged APOE4 carriers. Cortex. 2014 Aug;57:167-76. doi: 10.1016/j.cortex.2014.04.006. Epub 2014 Apr 30. PMID 24905971
- [Background] Sheline YI, Morris JC, Snyder AZ, Price JL, Yan Z, D'Angelo G, Liu C, Dixit S, Benzinger T, Fagan A, Goate A, Mintun MA. APOE4 allele disrupts resting state fMRI connectivity in the absence of amyloid plaques or decreased CSF Abeta42. J Neurosci. 2010 Dec 15;30(50):17035-40. doi: 10.1523/JNEUROSCI.3987-10.2010. PMID 21159973
- [Background] Koh MT, Haberman RP, Foti S, McCown TJ, Gallagher M. Treatment strategies targeting excess hippocampal activity benefit aged rats with cognitive impairment. Neuropsychopharmacology. 2010 Mar;35(4):1016-25. doi: 10.1038/npp.2009.207. Epub 2009 Dec 23. PMID 20032967
- [Background] Sanchez PE, Zhu L, Verret L, Vossel KA, Orr AG, Cirrito JR, Devidze N, Ho K, Yu GQ, Palop JJ, Mucke L. Levetiracetam suppresses neuronal network dysfunction and reverses synaptic and cognitive deficits in an Alzheimer's disease model. Proc Natl Acad Sci U S A. 2012 Oct 16;109(42):E2895-903. doi: 10.1073/pnas.1121081109. Epub 2012 Aug 6. PMID 22869752
- [Background] Devi L, Ohno M. Effects of levetiracetam, an antiepileptic drug, on memory impairments associated with aging and Alzheimer's disease in mice. Neurobiol Learn Mem. 2013 May;102:7-11. doi: 10.1016/j.nlm.2013.02.001. Epub 2013 Feb 13. PMID 23416036
- [Background] Bakker A, Krauss GL, Albert MS, Speck CL, Jones LR, Stark CE, Yassa MA, Bassett SS, Shelton AL, Gallagher M. Reduction of hippocampal hyperactivity improves cognition in amnestic mild cognitive impairment. Neuron. 2012 May 10;74(3):467-74. doi: 10.1016/j.neuron.2012.03.023. PMID 22578498
- [Background] Vossel KA, Beagle AJ, Rabinovici GD, Shu H, Lee SE, Naasan G, Hegde M, Cornes SB, Henry ML, Nelson AB, Seeley WW, Geschwind MD, Gorno-Tempini ML, Shih T, Kirsch HE, Garcia PA, Miller BL, Mucke L. Seizures and epileptiform activity in the early stages of Alzheimer disease. JAMA Neurol. 2013 Sep 1;70(9):1158-66. doi: 10.1001/jamaneurol.2013.136. PMID 23835471
- [Background] Palop JJ, Chin J, Roberson ED, Wang J, Thwin MT, Bien-Ly N, Yoo J, Ho KO, Yu GQ, Kreitzer A, Finkbeiner S, Noebels JL, Mucke L. Aberrant excitatory neuronal activity and compensatory remodeling of inhibitory hippocampal circuits in mouse models of Alzheimer's disease. Neuron. 2007 Sep 6;55(5):697-711. doi: 10.1016/j.neuron.2007.07.025. PMID 17785178
- [Background] Tuminello ER, Han SD. The apolipoprotein e antagonistic pleiotropy hypothesis: review and recommendations. Int J Alzheimers Dis. 2011 Feb 24;2011:726197. doi: 10.4061/2011/726197. PMID 21423560
- [Background] Dickerson BC, Salat DH, Bates JF, Atiya M, Killiany RJ, Greve DN, Dale AM, Stern CE, Blacker D, Albert MS, Sperling RA. Medial temporal lobe function and structure in mild cognitive impairment. Ann Neurol. 2004 Jul;56(1):27-35. doi: 10.1002/ana.20163. PMID 15236399
- [Background] Mohajeri MH, Saini K, Schultz JG, Wollmer MA, Hock C, Nitsch RM. Passive immunization against beta-amyloid peptide protects central nervous system (CNS) neurons from increased vulnerability associated with an Alzheimer's disease-causing mutation. J Biol Chem. 2002 Sep 6;277(36):33012-7. doi: 10.1074/jbc.M203193200. Epub 2002 Jun 14. PMID 12068009
- [Background] Tampellini D, Capetillo-Zarate E, Dumont M, Huang Z, Yu F, Lin MT, Gouras GK. Effects of synaptic modulation on beta-amyloid, synaptophysin, and memory performance in Alzheimer's disease transgenic mice. J Neurosci. 2010 Oct 27;30(43):14299-304. doi: 10.1523/JNEUROSCI.3383-10.2010. PMID 20980585

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AGB101 220 mg, Then Placebo | Placebo, Then AGB101 220 mg
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: One enrolled subject did not have detectable LEV in their blood sample and was discarded in analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | AGB101 220 mg, Then Placebo | Placebo, Then AGB101 220 mg | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Categorical [Count of Participants; unit: Participants] — Population: One enrolled subject did not have detectable LEV in their blood sample and was discarded in analysis
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 5 | 4 | 9
    >=65 years | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: One enrolled subject did not have detectable LEV in their blood sample and was discarded in analysis
  years | 66 (4) | 67 (5) | 66.2 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One enrolled subject did not have detectable LEV in their blood sample and was discarded in analysis
  Participants
    Female | 9 | 6 | 15
    Male | 4 | 6 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: One enrolled subject did not have detectable LEV in their blood sample and was discarded in analysis
  Participants
    Hispanic or Latino | 0 | 0 | 0
    Not Hispanic or Latino | 13 | 12 | 25
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: One enrolled subject did not have detectable LEV in their blood sample and was discarded in analysis
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 13 | 12 | 25
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Population: One enrolled subject did not have detectable LEV in their blood sample and was discarded in analysis
  participants
    United States | 13 | 12 | 26
Apolipoprotein E (APOE) Status [Count of Participants; unit: Participants] — Population: One enrolled subject did not have detectable LEV in their blood sample and was discarded in analysis
  Participants
    APOE e4 Carrier | 3 | 2 | 5
    APOE e4 Non-Carrier | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Functional Connectivity Strengths of Neural Networks
Description: The seed-based functional connectivity strengths of the hippocampus network and the default mode network will be employed to measure the changes between AGB101 and Placebo perturbation. The functional connectivity strengths will be measured with the median of the Pearson cross-correlation coefficients over entire brain regions.
Time Frame: 2 weeks after treatment between AGB101 and Placebo
Population: A total of 25 subjects who were treated with AGB 101 and Placebo (order-balanced), then conducted a paired t-test to detect the treatment effect vs placebo.
Measure: Median (Standard Deviation); unit: Pearson coefficient
Groups:
- AGB101 220 mg: AGB101 220 mg/day capsule, once daily dosing for 2 weeks.
  AGB101 220 mg: AGB101 oral dose of 220 mg/day capsule, given as once-daily dosing.
- Placebo: Placebo, given as a capsule, once daily for 2 weeks.
  Placebo: Placebo, oral capsule given once-daily.
Arm/Group | AGB101 220 mg | Placebo
Number analyzed (Participants) | 25 | 25
Pearson coefficient | 0.233 (0.132) | 0.318 (0.127)
Statistical Analysis 1: Comparison: AGB101 220 mg vs Placebo; The null hypothesis (H0) of this superiority trials asserts that there is no true difference in functional connectivity between the interventions of placebo and AGB101, and the alternative hypothesis (H1) states that there is a difference between the interventions of placebo and AGB101. A type I error is the error of rejecting H0 when it is actually true; Test type: Superiority; p = 0.007567, t-test, 2 sided; Median Difference (Final Values) = -0.083, 95% CI 2-sided [-0.0886 to -0.0774], Standard Deviation 0.0056

2. Secondary Outcome: Rey Auditory Verbal Learning Test (AVLT), Delayed Recall Scaled Integer. The Higher is the Better
Description: Rey Auditory Verbal Learning Test (AVLT), delayed recall Scaled integer will be employed to measure the episodic memory changes before and after AGB101 treatment. The AVLT score will be recorded as a standard score. The theoretical range: min 50, max 155, the higher the better. The higher the number is, the better the memory. It is an integer number.
Time Frame: Placebo vs AGB101 2 weeks after treatment paired t-test
Population: Measure RAVLT Delayed recall standard score memory test
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AGB101 220 mg | Placebo
Number analyzed (Participants) | 25 | 25
score on a scale | 108 (17) | 105 (16)
Statistical Analysis 1: Comparison: AGB101 220 mg vs Placebo; The null hypothesis (H0) of this trial asserts that there is no true difference in AVLT between the interventions of placebo and AGB101, and the alternative hypothesis (H1) states that there is a difference between the interventions of placebo and AGB101. A type I error is the error of rejecting H0 when it is actually true; Test type: Superiority; p = 0.900593, t-test, 2 sided; Mean Difference (Final Values) = 3.12, 95% CI 2-sided [1.72 to 4.52], Standard Deviation 1.40

ADVERSE EVENTS:
Time Frame: From Baseline Visit Through 4 Week Follow Up Call (an average of 12 weeks)
Groups:
- AGB101 220 mg: AEs judged related to intervention while on AGB101 220 mg
- Placebo: AEs judged related to intervention while on Placebo
Arm/Group | AGB101 220 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 6/26 | 3/26
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AGB101 220 mg (N=26) | Placebo (N=26)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Sleepiness (General disorders) | 1 (1) | 0 (0)
Brain Zaps (Nervous system disorders) | 0 (0) | 1 (1)
Visual Aura (Nervous system disorders) | 0 (0) | 1 (1)
Cold Symptoms (Infections and infestations) | 1 (1) | 0 (0)
Feeling Jittery (Nervous system disorders) | 1 (1) | 0 (0)
Depressed Mood (Psychiatric disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
26 total patients were enrolled in the project, and 25 total patients were included in analysis. One enrolled subject did not have detectable LEV in their blood sample and was discarded in analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is an agreement between Dr. Li and AgeneBio since AgeneBio supplies AGB101 drug to Dr. Li's for conducting the trial. The only restriction on the PI is that the sponsor can review results communications prior to public release.

DOCUMENTS (2):
  • Study Protocol (2019-04-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT03461861/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT03461861/SAP_002.pdf